CLINICAL TRIAL: NCT05176834
Title: Self-applied Photobiomodulation Therapy With a Home-use Device for the Prevention and/or Acceleration of Healing of Radiation-induced Oral Mucositis in Patients With Head and Neck Malignancies - A Feasibility Study
Brief Title: Photobiomodulation Home-use Device for Prevention or Treatment of Oral Mucositis in Patients With Head&Neck Malignancies
Acronym: PBM&OM-01
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Erika Carmel ltd (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 0183-21-RMB
Record Dates: First submitted 2021-12-13; First posted 2022-01-04 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Mucositis; Head and Neck Cancer; Radiotherapy Side Effect
MeSH Terms: conditions — Mucositis; Head and Neck Neoplasms; Radiation Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- B-Cure laser pro (Experimental): In case of appearance of mucositis, patients will receive standard treatment as usual (rinses, painkillers, etc.). In addition, study participants will treat themselves with the B-Cure laser pro before each radiation therapy session at the clinic and will continue with daily treatment until the disappearance of the mucositis should it develop.
  Interventions: Device: B-Cure laser pro

INTERVENTIONS:
Device: B-Cure laser pro — The B-Cure laser pro is a portal, non-invasive, photobiomodulation device, that emits light in the near infrared (808nm) over an area of 1X4.5 cm2 with power output of 250mW, and energy dose of 1J/cm2.

SUMMARY:
Patients with head and neck malignancy that are treated with Radiation Therapy [RT] are expected to develop Oral Mucositis (OM) in 60% of cases. Mucositis is a side effect of radiation and / or chemotherapy that causes severe pain and inability to eat and drink and a decrease in quality of life. In addition it may impair the treatment protocol and treatment outcomes.

Photobiomodulation is a non-ionizing optical radiation in the near or near-infrared range used for acceleration of wound healing and pain reduction. Photobiomodulation therapy for the reduction of mucositis is included in the International Guidelines of the MASCC / ISOO Association and the British NICE. To date the treatment has been performed by members of professional medical staff in hospitals or clinics.

The study device is home-used photobiomodulation device approved for indications of pain reduction and acceleration of wound healing. The device has shown efficacy in treating mucositis around dental implants in a clinical trial and after oncological treatments in a limited number of cases as reported in the scientific literature.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with malignant neoplasm in the oral cavity, pharynx or salivary glands.
2. The patient should receive a continuous course of radiation therapy (IMRT) with all of the following criteria applicable:

   * For a period of 3-7 weeks, 5-6 fractions per week.
   * A minimum cumulative dose of 30Gy expected to cause OM (ORAL MUCOSITIS) by the third week. Or: Based on the clinical judgment of the Radiation Oncologist and BED2 ≥ 30 Gy
   * The treatment field will include at least one oral site (buccal mucosa, floor of mouth, tongue, hard palate, retro-molar trigon, lips or oropharynx)
   * With or without chemotherapy and / or immunotherapy at the same time.
3. A patient with an ECOG PS functional status equal to or less than 2
4. Able to read and understand the informed consent form (ICF) and voluntarily provided informed consent
5. The patient is able to undergo intra-oral treatments
6. The patient is willing to perform the protocol.

Exclusion Criteria:

1. The patient underwent previous radiation to the current therapeutic field
2. The patient has health conditions of the teeth or mouth that will prevent the application of intra-oral treatment
3. The patient receives non-standard treatment for mucositis such as benzidamine, palifermin, etc.
4. The patient is enrolled to any other clinical trial that includes treatment or intervention that may affect the course of mucositis.
5. The patient has a diagnosis that affects the healing of wounds (eg diabetes, lupus, etc.)
6. Pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-01-31 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients performing at least 50% of expected daily treatments during radiotherapy period. | 7 weeks
  The patients are expected to treat themselves 5 times a week during the 7 week period of radiotherapy, accumulating to a total of 35 treatments. The date of each treatment will be documented in a diary. The number of treatment actually done divided by the 35 expected treatments will be calculated. The outcome is the proportion of patients that will treat themselves at least 18 treatments out of the 35 expected (at least 50%).

SECONDARY OUTCOMES:
The proportion of the patients that will experience severe oral mucositis | 7 weeks
  The proportion of the patients that will experience severe oral mucositis defined as grade 3 or 4 of the World Health Organization (WHO) grading for oral mucositis, according to the following:
  Grade 0=the patient has no signs and symptoms; Grade 1=painless ulcers, edema, or mild soreness; Grade 2=painful erythema, edema, or ulcers but able to eat; Grade 3=painful erythema, edema, or ulcers but unable eat; Grade 4=requires parenteral or enteral support

CONTACTS AND LOCATIONS:
Locations (1):
- Rambam Medical Center, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Salman S, Abdalla-Aslan R, Awawdi A, Tarabeih R, Billan S. From clinic to couch: a pilot study of home-use photobiomodulation for radiation-induced oral mucositis and dermatitis. Support Care Cancer. 2025 Nov 7;33(12):1023. doi: 10.1007/s00520-025-10037-3. PMID 41201561